CLINICAL TRIAL: NCT05425056
Title: A Phase 3, Prospective, Randomized, Multicenter, Single-blind, Controlled Study Evaluating Arteriovenous Fistula Outcomes With and Without a Perivascular Sirolimus Eluting Collagen Implant (The ACCESS 2 Trial)
Brief Title: A Study Testing the Use of a Perivascular Sirolimus Formulation (Sirogen) in ESRD Patients Undergoing AV Fistula Surgery
Acronym: ACCESS2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vascular Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: VT-305
Record Dates: First submitted 2022-06-10; First posted 2022-06-21 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2024-08

CONDITIONS: Complication of Renal Dialysis; End Stage Renal Disease; End Stage Kidney Disease; ESRD; Chronic Kidney Failure; Complication of Hemodialysis; Vascular Access Complication; Arteriovenous Fistula
Keywords: Arteriovenous Fistula; Hemodialysis vascular access; Dialysis fistula; Dialysis access
MeSH Terms: conditions — Kidney Failure, Chronic; Arteriovenous Fistula | interventions — Sirolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Experimental): Subjects randomized to the treatment arm will undergo AV fistula surgery and will receive the Sirolimus eluting Collagen Implant (SeCI).
  Interventions: Drug: Sirolimus
- Control Arm (No Intervention): Subjects randomized to the control arm will undergo AV fistula surgery alone and will not receive an implant.

INTERVENTIONS:
Drug: Sirolimus — SeCI placed at and around the site of the anastomosis of an AV fistula, immediately following completion of a successful AV fistula surgery.
  Other Names: Sirolimus-eluting Collagen Implant; SeCI; Sirogen
  Arms: Treatment Arm

SUMMARY:
The primary study objective is to evaluate the benefit of the Sirolimus eluting Collagen implant (SeCI; Sirogen), a single dose prophylactic treatment delivered intraoperatively at the time of surgical creation of an arteriovenous fistula for hemodialysis vascular access.

DETAILED DESCRIPTION:
This is a Phase 3, multicenter, randomized, single-blind, controlled, study designed to evaluate the efficacy and safety of the use of the Sirolimus-eluting Collagen Implant (SeCI) in subjects who are on hemodialysis and are undergoing surgical creation of an AV fistula in comparison to subjects who do not receive the implant.

Subjects of either gender, who are at least 65 years of age, undergoing hemodialysis, and require a new single stage radiocephalic end to side fistula will be eligible to participate in this study. Subjects who meet eligibility criteria and undergo successful AV fistula creation will be eligible for enrollment. The study plans to enroll approximately 120 subjects, randomized in a 1:1 ratio. Enrolled subjects will be followed for a period of one year from the time of their index surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years or older
* Currently on hemodialysis for ≤12 months
* Successful creation of a single stage radiocephalic end to side fistula

Exclusion Criteria:

* Prior AV access created on the limb where the fistula surgery is planned
* Planned start of peritoneal dialysis within 6 months of randomization
* Known hypersensitivity to the following: sirolimus, beef or bovine collagen
* Known to be HIV positive
* Prisoner, mentally incompetent, and/or current alcohol or drug abuser

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 136 (Actual)
Dates: Start 2022-08-26 (Actual); Primary Completion 2025-03-18 (Actual); Study Completion 2025-08-29 (Actual)

PRIMARY OUTCOMES:
Clinical Fistula Maturation (FM) | 6 Months
  Clinical Fistula Maturation (FM) is defined as a fistula that can be cannulated with 2-needles for at least 75% of the dialysis sessions, including 3 consecutive sessions with a mean Qb of 300 mL/min (unless the prescribed Qb is <300 mL/min) performed during any continuous 30 day period that commences no later than 180 days after randomization.
  The primary endpoint will be summarized as a time-to-event endpoint for the SeCI (Sirogen) and control groups by reporting the cumulative proportion of AVF that achieve FM over time [defined as the interval from access placement to the first session that the fistula can be cannulated with 2 needles (contributing to the FM definition)].

SECONDARY OUTCOMES:
Fistula Suitability for Dialysis at 12 months (FSD12) | 1 year
  Fistula Suitability for Dialysis at 12 months (FSD12) defined as a fistula that can be used for dialysis using 2 needles for at least 75% of the dialysis sessions performed during a 30 day period that commences on day 330.
Secondary Patency (SP) | 1 year
  Secondary Patency (SP) defined as the interval from the time of randomization until access abandonment.
Time To First Dialysis (TTFD) | 1 year
  Time To First Dialysis (TTFD) defined as the interval from the time of randomization to the first of three consecutive dialysis sessions using 2 needles with a mean Qb of ≥300 mL/min (unless the prescribed Qb is <300 mL/min).
Mature Fistula with Preserved Function at 12 Months (MFPF) | 1 year
  Mature Fistula with Preserved Function at 12 Months (MFPF) defined as a fistula that can be cannulated with 2 needles for at least 75% of the dialysis sessions, including 3 consecutive sessions with a mean Qb of ≥300 mL/min (unless the prescribed Qb is <300 mL/min) performed during any continuous 30-day period that commences no later than 180 days after randomization (i.e., fistula achieves FM) AND can be used for dialysis using 2-needles for at least 75% of the for the dialysis sessions performed during a 30-day period that commences on day 330 (FSD12).
Durable Fistula Maturation (DFM) | 1 year
  Durable Fistula Maturation (DFM) defined as a fistula that can be cannulated with 2 needles for at least 75% of the dialysis sessions, including 3 consecutive sessions with a mean Qb of ≥300 mL/min performed during any continuous 30-day period that commences no later than 180 days after randomization (i.e., fistula achieves FM) AND can be used for dialysis using 2-needles with a mean Qb of ≥300 mL/min for the dialysis sessions performed during a 30-day period that commences on day 330.
Cumulative Fistula Use (CFU) | 1 year
  Cumulative Fistula Use (CFU) defined as the number of dialysis sessions performed using the study fistula with 2 needles and a mean Qb of ≥300 mL/min. CFU is calculated from the time of fistula creation to the end of study period or upon reaching an intercurrent event (Fistula abandonment, Death, Transfer to PD or transplant) or is lost to follow up.
Cumulative Catheter Exposure (CCE) | 1 year
  Cumulative Catheter Exposure (CCE) is defined as the number of days a hemodialysis central venous catheter (CVC) is in situ and the duration of CVC exposure is calculated from the day of fistula creation (i.e., day of randomization) to the end of study period or upon reaching an intercurrent event.

CONTACTS AND LOCATIONS:
Overall Officials: Sriram Iyer, MD, Study Director — Vascular Therapies, Inc.
Locations (22):
- United States (17):
  - Veterans Affairs San Diego Health Center, San Diego, California
  - Lundquist Institute for Biomedical Innovation, Torrance, California
  - MedStar Cardiovascular Research Network at MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - American Access Care of Miami, Miami, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - University of Louisville, Louisville, Kentucky
  - The Brigham and Women's Hospital, Boston, Massachusetts
  - Mount Sinai Hospital, New York, New York
  - Atrium Health, Charlotte, North Carolina
  - Surgical Specialists of Charlotte, Charlotte, North Carolina
  - The Regional Medical Center/Dialysis Access Institute, Orangeburg, South Carolina
  - James Eric Gardner, MD PC, Memphis, Tennessee
  - Arteries & Veins, El Paso, Texas
  - Houston Methodist, Houston, Texas
  - Houston Methodist, Sugar Land, Texas
  - Sentara Norfolk General Hospital/Sentara Health Research Center, Norfolk, Virginia
- United Kingdom (5):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - St Helier Hospital, Carshalton
  - NHS Greater Glasgow and Clyde, Glasgow
  - Barts Health NHS Trust of Royal London Hospital, London
  - St George's University Hospitals NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) collected in this study will not be shared.